CLINICAL TRIAL: NCT06191042
Title: A Multicenter, Phase 1b, Double-blind, Placebo-controlled Study to Evaluate the Safety and Tolerability, and the Efficacy of Si-544 in Adults With Psoriasis Vulgaris or Psoriatic Arthritis
Brief Title: A Study to Evaluate the Safety and Tolerability, and the Efficacy of Si-544 in Adults With Psoriasis Vulgaris or Psoriatic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: selectION Therapeutics GmbH (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SEL-002; 2023-507393-40 (Other: EU CT Number)
Record Dates: First submitted 2023-12-10; First posted 2024-01-05 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Psoriasis Vulgaris; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- si-544 (Experimental)
  Interventions: Drug: si-544
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: si-544 — Subcutaneous injection in the abdomen
  Arms: si-544
Drug: Placebo — Subcutaneous injection in the abdomen
  Arms: Placebo

SUMMARY:
The main objective of this study is to investigate the safety and tolerability of si-544.

Other objectives are to study the metabolism of si-544 in the body and to assess the effects of si-544 on cells of the body's immune system (immune cells) that have been chronically activated by the disease. Likewise, the effect of si-544 on inflammatory responses in the body triggered by the disease and other disease symptoms will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the capacity for consenting, was informed about the nature, the scope, and the relevance of the clinical study, voluntarily agrees in participation and in the study provisions, and duly signed the ICF approved by the ethics committee before any study-related procedure is performed
2. Men and women aged ≥18 to 75 years
3. Willing and able to adhere to the protocol requirements
4. Women of childbearing potential must:

   1. have a negative pregnancy test (blood) at Screening and a negative pregnancy test (urine) at Day 1
   2. agree to use, and be able to comply with, highly effective measures of contraceptive control (failure rate less than 1% per year when used consistently and correctly) without interruption, from Screening through 30 days after the last IMP injection

   Reliable methods for this study are:

   i. combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal) ii. progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable) iii. intrauterine device iv. intrauterine hormone-releasing system v. bilateral tubal occlusion vi. vasectomized sexual partner (provided that the partner is the sole sexual partner of the woman of childbearing potential and has received medical assessment of the surgical success) vii. sexual abstinence (only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatment) Abstinence is only accepted as true abstinence: when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods and withdrawal] is not an acceptable method of contraception).

   c. agree to abstain from breast feeding during the study participation and for 90 days after the last IMP injection
5. Postmenopausal (no menses for at least 1 year without alternative medical cause) or surgically sterile women (tubal ligation, hysterectomy, or bilateral oophorectomy)
6. Men must agree to practice true abstinence or to use a condom during sexual contact with a pregnant woman or a woman of childbearing potential during study participation and for at least 90 days after the last IMP injection, even after undergoing a successful vasectomy.

   Ps-specific inclusion criteria:
7. Diagnosis of Ps at least 3 months before Screening
8. Active Ps with ≥3% BSA involved and with at least 1 psoriatic plaque (other than nail change)

PsA-specific inclusion criteria:

7. Diagnosis of PsA based on the classification for psoriatic arthritis criteria (CASPAR) at least 3 months before Screening

8. Diagnosis of active Ps with at least 1 psoriatic plaque (other than nail change)

9. Active PsA defined as

1. ≥1 tender joint out of 68 assessed joints, and
2. ≥1 swollen joint out of 66 assessed joints (dactylitis of a digit counts as one joint each), and
3. negative results for rheumatoid factor and anti-cyclic citrullinated peptide antibodies

Exclusion Criteria:

1. Known history of hypersensitivity to constituents or excipients in the pharmaceutical formulation of the IMP
2. Uncontrolled hypertension or uncontrolled diabetes, as judged by the investigator
3. Chronic disease other than Ps or PsA not adequately controlled by stable treatment (ie, no changes or initiation of treatment within 4 weeks before Screening and Day 1)
4. History of seizures
5. Presence or history of paresthesia or neuropathy
6. Clinically significant ECG abnormalities, as judged by the investigator
7. Clinically relevant disease which could affect the safety of the subject during the study or impede the subject's ability to complete the study, as assessed by the investigator
8. Presence of acute infection within 7 days before Screening or Day 1, as judged by the investigator
9. Known or active infection with Mycobacterium tuberculosis and/or positive tuberculosis interferon γ release assay result at Screening
10. Known or active infection with HIV, hepatitis B virus, or hepatitis C virus
11. Known or suspected abuse of alcohol, drugs, or medicinal products
12. Therapy with biologics used for the treatment of Ps and/o PsA (including those under investigation) within 1 year before Day 1
13. UV phototherapy or systemic therapy (except methotrexate for the treatment of PsA) within 4 weeks of Day 1
14. Vaccination within 2 weeks (for live vaccines within 4 weeks) before Day 1 and/or planned vaccination during the treatment period
15. Current or previous (within 4 weeks before Day 1) participation in another clinical study with an IMP or a medical device
16. Employee of the sponsor, or employee, or relative of the investigator
17. Committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
18. Legal incapacity or limited legal capacity

    Ps-specific exclusion criteria:
19. Drug-induced psoriasis

PsA-specific exclusion criteria:

19. Late stage PsA with deformed joints

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Determination of safety and tolerability of treatment with si-544 | From Day -35 to Day 106
  Occurrence of adverse events (AEs) and serious AEs (SAEs), including description of type, frequency, severity, and causal relationship of adverse events (AEs) and serious AEs
Determination of safety and tolerability of treatment with si-544 | From Day 1 (Baseline) to Day 106
  Change in clinical laboratory, electrocardiogram (ECG), vital signs, and peripheral oxygen saturation from Baseline to all assessed timepoints

SECONDARY OUTCOMES:
Determination of the plasma concentrations of free si-544 | Day 1 (Baseline) and Day 25
  Plasma concentrations of free si-544
Determination of the pharmacodynamics (PD) of si-544 as assessed by the number of T cells in peripheral blood | From Day 1 (Baseline) to Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the number of T cells in peripheral blood
Determination of the pharmacodynamics (PD) of si-544 as assessed by immunophenotypes of T cell subsets | From Day 1 (Baseline) to Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in immunophenotypes of T cell subsets
Determination of the pharmacodynamics (PD) of si-544 as assessed by serum cytokine levels | From Day 1 (Baseline) to Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in serum cytokine levels
Determination of the immunogenicity of si-544 treatment | From Day 1 (Baseline) to Day 29 (Week 5) and Week 16
  Change in anti-drug antibodies against si-544 in serum
Determination of the efficacy of si-544 treatment as assessed by psoriasis area and severity index (PASI) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the psoriasis area and severity index (PASI)
Determination of the efficacy of si-544 treatment as assessed by psoriasis area and severity index (PASI) response rate | At Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Difference in psoriasis area and severity index (PASI) response rate (defined as subjects with ≥1 score improvement from Baseline)
Determination of the efficacy of si-544 treatment as assessed by physician's global assessment (PGA) of disease activity | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the physician's global assessment (PGA) of disease activity
Determination of the efficacy of si-544 treatment as assessed by body surface area (BSA) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in affected body surface area (BSA)
Determination of the efficacy of si-544 treatment as assessed by a numeric rating scale (NRS) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the mean itch using a numeric rating scale (NRS)
Determination of the efficacy of si-544 treatment as assessed by a numeric rating scale (NRS) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the worst itch using a numeric rating scale (NRS)
Determination of the efficacy of si-544 treatment on symptoms of psoriasis vulgaris (Ps) in Ps patients only as assessed by dermatological life quality index (DLQI) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the dermatological life quality index (DLQI)
Determination of the efficacy of si-544 treatment on symptoms of psoriatic arthritis (PsA) in PsA patients only as assessed by psoriatic arthritis quality of life (PsAQoL) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the psoriatic arthritis quality of life (PsAQoL)
Determination of the efficacy of si-544 treatment on symptoms of psoriatic arthritis (PsA) in PsA patients only (assessment of pain) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the subject's assessment of pain using a visual analog scale (VAS)
Determination of the efficacy of si-544 treatment on symptoms of psoriatic arthritis (PsA) in PsA patients only as assesses by the 66 swollen joint count (SJC66) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the 66 swollen joint count (SJC66)
Determination of the efficacy of si-544 treatment on symptoms of psoriatic arthritis (PsA) in PsA patients only as assessed by the 68 tender joint count (TJC68) | From Day 1 (Baseline) to Day 15, Day 29 (Week 5), Week 8, Week 12 and Week 16
  Change in the 68 tender joint count (TJC68)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Klostermann, Dr., Study Director — selectION Therapeutics GmbH
Locations (4):
- Germany (4):
  - selectION Clinical Trial Site, Bad Bentheim
  - selectION Clinical Trial Site, Berlin
  - selectION Clinical Trial Site, Blankenfelde-Mahlow
  - selectION Clinical Trial Site, Hamburg

IPD SHARING:
Plan to Share IPD: No
Due to uncertainties in EU data protection legislation individual deidentified participant data are not shared. The main uncertainty is the concept of what "deidentified" means. It appears not to mean that the data set of a person is simply separated from the person's name. What additional operations have to be done appears to depend on technological capabilities to re-identify the persons associated with the data set. A common perception is that the technological capabilities for re-identification are permanently increasing. This could have the effect that public data sets that are regarded as deidentified now might become re-identifiable data sets in the future. Once this happens, the sponsor is no longer able to make the publication of the data sets un-happen. This could result in sanctioning by EU data protection authorities. The sponsor wants to avoid this.